CLINICAL TRIAL: NCT03885128
Title: Intra Versus Extra-thoracic Oscillations in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed El-Moatasem Mohamed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/001741
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vest arm (Experimental): high frequency chest wall oscillation vest performed 4 times per week for 6 successive weeks for 30 patients
  Interventions: Device: High frequency extra thoracic oscillations vest
- Quake arm (Experimental): Vibratory positive expiratory pressure quake performed 4 times per week for 6 successive weeks for 30 patients
  Interventions: Device: Intrathoracic oscillatory quake

INTERVENTIONS:
Device: High frequency extra thoracic oscillations vest — Oscillations applied extra thoracic through vest device aiming for airway clearance
  Arms: Vest arm
Device: Intrathoracic oscillatory quake — Oscillation introduced intrathoracic through quake device through placing quake in mouth and ordering patient to breathing to move secretions
  Arms: Quake arm

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is the fourth-leading cause of death. It is a progressive illness that requires life-long treatment.Promoting airway clearance (AC) using mucolytics together with airway clearance techniques (ACTs) form the basis for pulmonary therapy in COPD care.Therefore, new airway clearance modalities are required to decrease the detrimental effects of accumulated secretions in COPD.

One of the devices used in AC is the high frequency chest wall oscillation (The Vest). HFCWO involves the use of an inflatable vest/jacket that covers the chest and is attached to an air pulse-generating compressor which rapidly inflates and deflates the vest, producing oscillations to the chest wall of 5-25 Hz.

Another new airway clearance modality is oscillating positive expiratory pressure(Quake) which combines PEP therapy with high frequency oscillations.

DETAILED DESCRIPTION:
The present study aimed to evaluate the effectiveness of the extra thoracic oscillations via high frequency chest wall oscillation vest (HFCWO) versus the intra thoracic oscillations via oscillatory positive expiratory pressure (OPEP) Quake device in COPD Group A: consists of 30 patients will be treated by high frequency chest wall oscillation vest along with their prescribed medical treatment. This program will be performed 4 times per week for 6 successive weeks.

Group B: consists of 30 patients will be treated by vibratory PEP (The Quake) along with their prescribed medical treatment. This program will be performed 4 times per week for 6 successive weeks.

ELIGIBILITY:
Inclusion Criteria:

* • All patients were diagnosed by chest physician based on the modified criteria defined in the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines 2017.

  * All patients were diagnosed as COPD for at least two years.
  * All Patients must use their prescribed medications.

Exclusion Criteria:

* All patients that had one of the following were excluded from the study. History of osteoporosis, significant gastro-esophageal reflux, hiatus hernia. Recent acute cardiac event (6 weeks) or congestive cardiac failure. Any significant musculoskeletal disorders. Presence of active hemoptysis Presence of malignant disease

Ages: 45 Years to 72 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Pulmonary function test (spirometry) | Before and 6 weeks
  * it measure ventilatory functions.
  * Then the patients sat comfortably and upright while putting the nose clip and relax.
  * The patient was asked to inhale as deeply as possible, hold the breath, and then inserted the mouthpiece carefully into the mouth.
  * The patient held the mouthpiece tightly between the lips, and kept tongue down.
  * The patient was asked to exhale for as long as possible and blow for at least 6 seconds.

SECONDARY OUTCOMES:
impulse oscillometry | before and 6 weeks
  The patient was in sitting position, Legs kept uncrossed The patient firmly supported his cheeks during measurement. The mouthpiece was at a comfortable height so that the neck is slightly extended and ensure that there is a tight seal between the mouthpiece and lips to prevent air leak.
  The patient was instructed to perform normal tidal breathing in a relaxed state during the procedure.
  The recording was performed for at least 30-45 s. During this period, around 120-150 sound impulses were pushed into the lungs from which the mean reactance and resistance values were determined at frequencies from 5 to 20 Hz.

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa M Badr, Professor, Study Chair — Professor physical therapy at Cairo university
Locations (1):
- Faculty of physical therapy, Dokki, Giza Governorate, Egypt